CLINICAL TRIAL: NCT07255118
Title: Effect of Music Intervention on Anxiety and Pain After Anatomical Endoscopic Enucleation of the Prostate: A Prospective Randomized Controlled Trial
Brief Title: Music Intervention During AEEP: A Prospective Randomized Controlled Trial
Acronym: AEEP-MUSIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: İrfan Şafak Barlas (Other)
Responsible Party: Sponsor-Investigator, İrfan Şafak Barlas, Urology Specialist, MD, FEBU, Acibadem University
Organization: Acibadem University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-10/425
Record Dates: First submitted 2025-11-20; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-01

CONDITIONS: Benign Prostatic Hyperplasia; Anxiety; Postoperative Pain Management
Keywords: AEEP; Music type; Postopertive comfort; State Anxiety Inventory; Visual Analog Scale
MeSH Terms: conditions — Prostatic Hyperplasia; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to one of two parallel groups: a music intervention group receiving perioperative music listening via headphones, and a control group receiving standard perioperative care without music. Each participant received only the intervention allocated to his assigned group, and outcomes were compared between the two independent groups.
Masking Description: This is an open-label study. No parties were masked because the nature of the music intervention made blinding infeasible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Group (Experimental): Participants undergoing AEEP who listened to standardized relaxing instrumental music via headphones during the perioperative period.
  Interventions: Behavioral: Music intervention
- Control Group (No Music) (No Intervention): Participants undergoing AEEP who received standard perioperative care without exposure to music.

INTERVENTIONS:
Behavioral: Music intervention — Patients listened to relaxing instrumental music beginning immediately before anesthesia induction and continuing throughout the procedure.
  Arms: Music Group

SUMMARY:
This prospective randomized controlled study investigates the effect of perioperative music listening on anxiety and postoperative pain in patients undergoing Anatomical Endoscopic Enucleation of the Prostate (AEEP) for benign prostatic hyperplasia. A total of 135 patients were randomized into two parallel groups: 67 patients listened to relaxing instrumental music during the perioperative period, while 68 patients received standard care without music. Anxiety was assessed using the State Anxiety Inventory (SAI) immediately before surgery and 2 hours postoperatively, and pain was evaluated using the Visual Analog Scale (VAS) at the postoperative 2nd hour. The study aims to determine whether a simple, non-pharmacological behavioral intervention can improve perioperative patient comfort and recovery outcomes in endoscopic prostate surgery.

DETAILED DESCRIPTION:
Benign prostatic hyperplasia (BPH) is one of the most common urological conditions in aging men, often requiring surgical intervention when medical therapy fails. Anatomical Endoscopic Enucleation of the Prostate (AEEP) has emerged as an effective and tissue-preserving surgical approach for managing BPH. Despite the minimally invasive nature of AEEP, perioperative anxiety and postoperative pain remain important determinants of patient comfort, satisfaction, and overall recovery.

Music listening is a simple, inexpensive, and non-pharmacological behavioral intervention that has been shown in various surgical disciplines to reduce anxiety, modulate pain perception, and improve patient experience. However, its potential benefits during AEEP have not been previously explored.

In this prospective randomized controlled trial, we evaluated the effect of perioperative music exposure on anxiety and acute postoperative pain among patients undergoing AEEP. A total of 135 male patients scheduled for AEEP were enrolled and randomized into two groups:

Music Group (n = 67): Patients listened to standardized relaxing instrumental music via headphones starting immediately before anesthesia induction and continuing during the procedure.

Control Group (n = 68): Patients received routine perioperative care without exposure to music.

Perioperative anxiety was measured using the State Anxiety Inventory (SAI) at two predefined time points: immediately before surgery and at the postoperative 2nd hour. Postoperative pain intensity was assessed using the Visual Analog Scale (VAS) 2 hours after the procedure. All surgical and anesthetic techniques were standardized across groups to minimize variability.

This study aims to determine whether perioperative music listening can serve as an effective adjunctive intervention to improve psychological well-being and reduce pain in patients undergoing AEEP. Findings from this research may support the integration of music into perioperative care pathways, offering a safe and easily applicable strategy to enhance patient-centered outcomes in endoscopic prostate surgery.

ELIGIBILITY:
Inclusion Criteria:

* male patients aged ≥40 years
* patients who underwent surgery under regional anesthesia without sedation
* patients who did not benefit from medical treatment for BPO
* preoperative International Prostate Symptom Score (IPSS) >19
* preoperative maximum urine flow rate (Qmax) <15 mL/sec
* post-voiding residual volume (PVR) >50 mL.

Exclusion Criteria:

* patients with urethral stricture
* patients who underwent urological treatments other than laser enucleation of the prostate
* patients with urinary tract infections and/or hematuria
* patients with urinary system malignancy
* patients with a history of previous prostate surgery
* patients with neurogenic bladder
* patients with hearing impairment
* patients with psychiatric disorders or those using medications prescribed by a psychiatrist.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Change in State Anxiety Inventory (SAI) Score | From baseline (immediately before surgery) to postoperative 2nd hour.
  Perioperative anxiety will be measured using the State Anxiety Inventory (SAI) at two time points: immediately before surgery (baseline) and at 2 hours postoperatively. The outcome represents the change in SAI score between these two assessments.

SECONDARY OUTCOMES:
Postoperative Pain Score Assessed by Visual Analog Scale (VAS) | Postoperative 2nd hour.
  Pain intensity will be evaluated using a 0-10 Visual Analog Scale (VAS) at the postoperative 2nd hour.

CONTACTS AND LOCATIONS:
Overall Officials: Irfan Safak Barlas, Urology Specialist, Principal Investigator — Acibadem Ankara Hospital
Locations (1):
- Acibadem Ankara Hospital, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the study is single-center, minimal-risk, and the dataset contains sensitive clinical information that cannot be fully de-identified in a reliable manner.